CLINICAL TRIAL: NCT06277349
Title: Multifocal-toric IOL Compared to Multifocal IOL Combined With Limbal Relaxing Incisions for Correction of Moderate Astigmatism During Cataract Surgery: A Randomised Trial
Brief Title: Multifocal-toric IOL Compared to Multifocal IOL Combined With Limbal Relaxing Incisions for Correction of Moderate Astigmatism During Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAUV1005
Record Dates: First submitted 2024-02-14; First posted 2024-02-26 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cornea; Astigmatism; Cataract
Keywords: multifocal; IOL; astigmatism; incision; cataract surgery; implant
MeSH Terms: conditions — Corneal Diseases; Astigmatism; Cataract; Surgical Wound

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with intra-patient comparison (bilateral study), patients are either receiving implant of a multifocal toric IOL or implant of a standard multifocal IOL combined with limbal relaxing incisions.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non toric multifocal IOL combined with corneal incisional surgery (Other): Non-toric Multifocal IOL (Rayner) - Model M-Flex 630F - CE marked since 2006 (in routine use). Surgery is performed under topical anaesthesia. Preoperatively, the horizontal meridian will be marked in the sitting position with a blue marking pen or insulin syringe at the limbus. The temporal self sealing incision, injection of viscoelastic substance, capsulorhexis, phacoemulsification, irrigation/aspiration of cortical material and injection of viscoelastic substance into the capsular bag are performed as standard procedure. Corneal limbal relaxing incisions (LRI) according to the Donnenefeld nomogram will be performed combined with standard non-toric multifocal IOL.
  Interventions: Device: Non-toric multifocal IOL
- Toric multifocal IOL alone (Other): Toric Multifocal IOL (Rayner) - Model M-Flex T 588 or 638 - CE marked since January 2007. Surgery is performed under topical anaesthesia. Preoperatively, the horizontal meridian will be marked in the sitting position with a blue marking pen or insulin syringe at the limbus. The temporal self sealing incision, injection of viscoelastic substance, capsulorhexis, phacoemulsification, irrigation/aspiration of cortical material and injection of viscoelastic substance into the capsular bag are performed as standard procedure. The multifocal toric IOL will be implanted.
  Interventions: Device: Toric multifocal IOL

INTERVENTIONS:
Device: Toric multifocal IOL — Implant of Multifocal toric intraocular lens only
  Other Names: Toric Multifocal IOL (Rayner) - Model M-Flex T 588 or 638 - CE marked since January 2007
  Arms: Toric multifocal IOL alone
Device: Non-toric multifocal IOL — Implant of non-toric multifocal lens plus incisional surgery
  Other Names: Non-toric Multifocal IOL (Rayner) - Model M-Flex 630F - CE marked since 2006 (in routine use)
  Arms: Non toric multifocal IOL combined with corneal incisional surgery

SUMMARY:
The purpose of the present study is to compare the outcome of multifocal toric intraocular lens with standard multifocal lens plus incisional surgery in patients undergoing bilateral cataract surgery.

DETAILED DESCRIPTION:
This is a randomized controlled trial with intra-patient comparison, 60 eyes (30 patients) with cataract and corneal astigmatism of 1.00 to 2.50 D (doctrine) took part in the trial. The trial assessed the efficacy of multifocal IOL (intraocular lens) with corneal pre-existing astigmatism and compare the outcomes of a multifocal toric IOL or a standard multifocal IOL combined with limbal relaxing incisions.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract and be planning to have both eyes operated on.
* Age 21 and older
* Have cataracts that allow IOL master biometry
* Regular corneal astigmatism 1.00 up to 2.50 D
* Difference of corneal astigmatism in both eyes to be equal to or less than 0.75D
* written informed consent to surgery and participation in the study
* Speak English

Exclusion Criteria:

* Relevant other ophthalmic diseases such as: pseudoexfoliation, glaucoma, traumatic cataract corneal scars, and other co-morbidity that could affect capsule bag stability ( e.g. Marfan syndrome)
* Irregular corneal astigmatism on Pentacam topography

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03-04 (Actual); Primary Completion 2011-01-04 (Actual); Study Completion 2011-01-04 (Actual)

PRIMARY OUTCOMES:
Composite scoring of unaided distance and near vision (monocularly) | 3 months
  Measurement of uncorrected and best corrected visual acuity will be done using a back-lit EDTRS chart placed at 4m.
  Near and distance unaided and corrected visual acuity will be measured, measuring reading speed, reading acuity and critical print size monocularly (Salzburg Reading Desk) and contrast vision under photopic and mesopic conditions (Pelli-Robson Chart).
  Reading speed, reading acuity and critical print size monocularly (Salzburg Reading Desk). The Salzburg Reading Desk (SRD) is the prototype of a reading chart that measures reading speed and reading distance. Contrast and light conditions are preset and reading distance (+/- 0.2 cm), reading speed and their changes during the examination are measured. This ensures an objective evaluation of measurements under the same conditions at every follow-up.
Residual astigmatism evaluation by Subjective Refraction and autorefraction (Topcon) | 3 months
  Measurement of residual astigmatism will be derived from autorefraction with an autorefractor (Topcon) with mean reading of 5 consecutive measurements in IOL mode, a subjective refraction by an optometrist using trial lenses and the cross cylinder method. All these measurements are non-invasive, non-contact and readily used in daily clinical practice.

DOCUMENTS (1):
  • Study Protocol (2009-02-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT06277349/Prot_000.pdf